CLINICAL TRIAL: NCT04153734
Title: Pembrolizumab + Platinum Doublets Without Radiation for Patients With PD-L1 ≥50% Locally Advanced Non-small Cell Lung Cancer: a Multicenter Prospective Single Arm Phase II Study
Brief Title: Pembrolizumab + Platinum Doublets Without Radiation for Programmed Death-ligand 1 (PD-L1) ≥50% Locally Advanced NSCLC
Acronym: Evolution
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kobe Minimally Invasive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Akito Hata, Akito Hata, Director of Division of Thoracic Oncology, Kobe Minimally Invasive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 57924-01
Record Dates: First submitted 2019-10-28; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer
Keywords: Pembrolizumab; Platinum doublets; Non-small cell lung cancer; Without radiation; Locally advanced; PD-L1 ≥50%
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Immunotherapy plus chemotherapy (Experimental): Combination of CDDP at 75 mg/m2 (day 1) or CBDCA at Area Under the Curve=6 (AUC=6) (day 1) + PEM at 500 mg/m2 (day 1) will be administered to patients with non-squamous cell carcinoma at 3-week intervals. To those with squamous cell carcinoma, CBDCA at AUC=6 (day 1) + nab-PTX at 100 mg/m2 (days 1, 8, and 15) will be administered at 3-week intervals. If there is no progression after the 4th course of induction therapy, it will be switched to maintenance therapy. For maintenance therapy, the combination of PEM at 500 mg/m2 (day 1) + Pembrolizumab at 200 mg (day 1) will be administered to patients with non-squamous cell carcinoma at 3-week intervals. To those with squamous cell carcinoma, Pembrolizumab at 200 mg (day 1) will be administered at 3-week intervals until disease progression or intolerable toxicity. Pembrolizumab administration should be continued for 2 years involving induction and maintenance therapies or until the 35th course.
  Interventions: Drug: Pembrolizumab; Drug: Cis Platinum; Drug: Carboplatin; Drug: Pemetrexed; Drug: nab paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab at 200 mg (day 1) will be administered to patients with non-squamous cell carcinoma at 3-week intervals. To those with squamous cell carcinoma, Pembrolizumab at 200 mg (day 1) will be administered at 3-week intervals until disease progression or intolerable toxicity. Pembrolizumab administration should be continued for 2 years involving induction and maintenance therapies or until the 35th course.
  Other Names: Keytruda
Drug: Cis Platinum — In patients with non-squamous histology, cisplatin (75 mg/m2) will be administered every 3 weeks until 4 cycles with pemetrexed and pembrolizumab.
  Other Names: CDDP
Drug: Carboplatin — In cisplatin-intolerable patients, carboplatin (AUC=6) will be administered every 3 weeks until 4 cycles with pemetrexed and pembrolizumab.
  Other Names: CBDCA
Drug: Pemetrexed — In patients with non-squamous histology, pemetrexed (500 mg/m2) will be administered every 3 weeks until progression or 2 years after initiation (35 cycles) with pembrolizumab.
  Other Names: Alimta
Drug: nab paclitaxel — In patients with squamous histology, nab-paclitaxel (100 mg/m2, day 1, 8, 15, tri-weekly) will be administered until 4 cycles with pembrolizumab.
  Other Names: Abraxane

SUMMARY:
This is a phase II, multicenter, single-arm, non-blind study. To 21 patients with PD-L1 ≥50% locally advanced non-small cell lung cancer, the combination of Pembrolizumab and platinum-doublets will be intravenously administered without radiotherapy to evaluate the efficacy and safety of combination therapy with Pembrolizumab and platinum-doublets.

DETAILED DESCRIPTION:
Trial procedure:

As induction therapy, ≤4 courses of combination therapy with Pembrolizumab at 200 mg (day 1) and a platinum preparation will be performed at 3-week intervals until disease exacerbation or intolerable toxicity appearance. Concerning combination therapy with a platinum preparation, the combination of cisplatin (CDDP) at 75 mg/m2 (day 1) or carboplatin (CBDCA) at Area Under the Curve=6 (AUC=6) (day 1) + pemetrexed (PEM) at 500 mg/m2 (day 1) will be administered to patients with non-squamous cell carcinoma at 3-week intervals. To those with squamous cell carcinoma, carboplatin (CBDCA) at AUC=6 (day 1) + nanoparticle albumin-bound paclitaxel (nab-PTX) at 100 mg/m2 (days 1, 8, and 15) will be administered at 3-week intervals. If there is no exacerbation after the 4th course of induction therapy, it will be switched to maintenance therapy. For maintenance therapy, the combination of PEM at 500 mg/m2 (day 1) + Pembrolizumab at 200 mg (day 1) will be administered to patients with non-squamous cell carcinoma at 3-week intervals. To those with squamous cell carcinoma, Pembrolizumab at 200 mg (day 1) will be administered at 3-week intervals until disease exacerbation or intolerable toxicity appearance. Pembrolizumab administration should be continued for 2 years involving induction and maintenance therapies or until the 35th course.

In each patient, diagnostic imaging will be performed every 6 weeks (42 ± 7 days)(every 9 weeks after Week 18, every 12 weeks after Week 45) to evaluate tumor-reducing effects. Using images, the response rate (RR) and progression-free survival (PFS) will be evaluated based on the "Guidelines for evaluating the treatment response of solid cancer (RECIST 1.1)". It is possible to continue treatment until PD evaluated by the attending physician based on the RECIST 1.1, intolerable toxicity appearance, the appearance of concomitant diseases affecting the continuation of treatment, discontinuation based on the study investigator's evaluation, withdrawal, pregnancy, incompliance with investigational-drug administration or procedures described in the protocol, appearance of management-related reasons, or completion of Pembrolizumab administration for 2 years involving induction and maintenance therapies or the 35th course. Even after PD is definitively diagnosed by the study investigator based on the RECIST 1.1, it is possible to continue treatment if the patient's condition is stable and if treatment is considered to be advantageous for the patient by the study investigator. During the trial period, adverse events should be examined,and severity grading should be performed according to the CTCAE（NCI Common Terminology Criteria for Adverse Events）version 5.0.

In cases without any response at first radiographic evaluation (6 weeks), local salvage therapy using radiotherapy is recommended by a discretion of doctors in charge. At that timing, such cases are treated as a censored case.

After enrollment of 10 cases, the trial will be early terminated by confirmed PD according RECIST at their initial radiographic evaluation (6 weeks) more than 3 cases.

Background:

Lung cancer accounts for 13% of all cancer patients. In 2012, 1,800,000 persons were newly diagnosed with lung cancer. Internationally, the number of patients who died of lung cancer in 2012 reached 1,600,000. Lung cancer is the most frequent cause of cancer-related death in males and the second most frequent cause of cancer-related death in females. Non-small cell lung cancer accounts for approximately 85% of all lung cancer lesions.

Concerning the treatment of non-small cell lung cancer, tumorectomy is performed in a stage in which radical resection is possible, and cure may be achieved at a relatively high probability. When radical resection is impossible, therapeutic strategies differ between patients with locally advanced cancer and those with remote metastasis. Standard treatment for stage III (locally advanced stage in which radical resection is impossible) non-small cell lung cancer is chemoradiotherapy (CRT). In some patients, radical cure may be achieved, but severe irreversible toxicities, such as treatment-associated death, pneumonia, and esophageal stenosis, may appear. In two phase III clinical studies regarding CRT for stage III lung cancer in which radical resection is impossible in Japan (WJTOG0105 and Osaka Lung Cancer Study Group 0007 studies), treatment-associated death and grade ≥3 pneumonia were observed in 3/4% and 2/10%, respectively. A recent phase II comparative clinical study in Japan (WJOG5008L study) compared CDDP + S-1 therapy with CDDP + vinorelbine therapy, and indicated that the treatment-associated mortality rates and incidences of grade ≥3 pneumonia were7.4/9.3% and 9.3/7.4%, respectively.

The rate at which radical cure was achieved by CRT was estimated to be approximately 20% based on the results of previous phase III clinical studies. In these studies, the PFS curve after CRT reached a plateau after 2 years. Briefly, if there is no relapse >2 years after treatment, the possibility of relapse-free survival may be high. This suggests that the 2-year PFS rate, which is also adopted as a primary endpoint in this study, is a surrogate marker of overall survival (OS).

Recently, the results of CRT in stage III patients in whom radical resection is impossible have not markedly improved, but it was demonstrated that additional immunotherapy after CRT prolonged the prognosis. A phase III comparative clinical study published in 2017 (PACIFIC study) indicated that the additional administration of a PD-L1 antibody, Durvalumab, to patients after CRT in stage III, in which radical resection is impossible, for 1 year prolonged the PFS (median: 16.8 vs. 5.6 months, respectively; HR 0.52; p<0.0001) and OS (median: not reached vs. 28.7 months, respectively; HR 0.68; p=0.0025) in comparison with a placebo. Based on the results of the study, 1-year Durvalumab administration following CRT was established as standard treatment for stage III cancer, which is impossible to treat by radical resection.

However, in the above study, randomization was performed after CRT, and the subjects did not include those with PD during CRT, those with grade ≥2 pneumonia, those with a reduction in the performance status (PS), those in whom CRT could not be completed, or those in whom Durvalumab could not be introduced within 42 days after CRT; Durvalumab should be additionally administered to patients who completed CRT, but it is difficult to notice treatment options before CRT. Furthermore, the results of the PACIFIC study may have been obtained, excluding these patients with poor prognoses.

In patients with PD-L1 ≥50% stage IV non-small cell lung cancer, the marked therapeutic effects of monotherapy with Pembrolizumab have been reported. In a phase III comparative study (Keynote-024), monotherapy with Pembrolizumab significantly prolonged the PFS (median: 10.7 vs. 6.7 months, respectively; HR 0.50; p<0.001) and OS (median: non-reached vs. non-reached, respectively; HR 0.60; p=0.005) in comparison with combination therapy with a platinum preparation, as primary treatment, in patients with PD-L1 ≥50% stage IV non-small cell lung cancer. Based on the results of the study, monotherapy with Pembrolizumab was established as primary standard treatment for PD-L1 ≥50% stage IV non-small cell lung cancer. In addition, a strategy to combine immunotherapy with chemotherapy was examined. A phase II comparative study involving patients with stage IV non-squamous, non-small cell lung cancer (Keynote-021 cohort G) showed that CBDCA + PEM + Pembrolizumab therapy prolonged the PFS (median: 19.0 vs. 8.9 months, respectively; HR 0.54; p=0.0067) and OS (median: non-reached vs. 20.9 months, respectively; HR 0.59; p=0.03) in comparison with CBDCA + PEM therapy. Interestingly, a population in which a plateau was reached after ≥24 months accounted for approximately 45% regardless of PD-L1. Furthermore, 16 of 20 PD-L1 ≥50% patients responded to treatment, with a response rate of 80%. Grades 3-5 adverse events occurred in 39.0% of the patients. There was a treatment-associated death (1.7%). To confirm the data, a phase III comparative study (Keynote-189) was conducted, supporting the efficacy of CBDCA + PEM + Pembrolizumab therapy. In the study, the response rate (61.4 vs. 22.9%, respectively), PFS (HR 0.36), and OS (HR 0.42) were significantly higher/longer in the 3-drug combination group (involving immunotherapy) among PD-L1 ≥50% patients. As the observation period was insufficient, it is difficult to evaluate the 2-year PFS and OS rates in the PD-L1 ≥50% patients, but the PFS and OS rates at 18 months were estimated to be approximately 40 and 70%, respectively, based on the survival curves. Concerning adverse events, the incidence of grade ≥3 toxicities and treatment-associated mortality rate in the 3-drug combination group were 67.2 and 6.7%, respectively, being slightly high. However, in the placebo group, the percentages were 65.8 and 5.9%, respectively; there were no differences. Furthermore, a phase III randomized controlled study of initial treatment for stage IV squamous cell carcinoma of the lung (Keynote-407) demonstrated the additive effects of pembrolizumab on combination therapy with a platinum preparation (CBDCA + nab-PTX). This therapy improved the response rate (58.4 vs. 38.0%, respectively), PFS (median: 6.4 vs. 4.8 months, respectively; HR 0.56; p<0.001), and OS (median: 15.9 vs. 11.3 months, respectively; HR 0.64; p=0.008). As the observation period was insufficient, it is difficult to evaluate the 2-year PFS and OS rates. However, the PFS and OS rates at 15 months were estimated to be approximately 30 and 50%, respectively, based on the survival curves. The hazard ratios (HRs) of PFS and OS in PD-L1 ≥50% patients were 0.37 and 0.64, respectively. Furthermore, there was no difference in the incidence of serious adverse events (grade ≥3) (69.8 vs. 68.2%, respectively). These data suggest the potent therapeutic effects of chemotherapy + Pembrolizumab in both PD-L1 ≥50% non-squamous and squamous cell carcinoma patients.

With respect to the effects of immunotherapy in an earlier stage, the efficacy of nivolumab as stage II/III preoperative therapy was reported. According to this report, nivolumab administered twice before surgery led to a major pathologic response (MPR rate: the rate of viable cells, <10%) in 9 (43%) of 21 patients. A higher MPR rate may be achieved by preoperative chemotherapy + immunotherapy. According to a report from the American Society of Clinical Oncology in 2018, the MPR rate after CBDCA + nab-PTX + Atezolizumab therapy (n=14), as stage II/III preoperative treatment, was 50%. In addition, at a meeting held by the World Conference on Lung Cancer in 2018, it was reported that pathological complete remission was achieved in 18 (60%) of 30 surgically treated patients after CBDCA + PTX + nivolumab therapy, and that an MPR was achieved in 6 (20%); the MPR rate was 80%. These data also suggest that immunotherapy is more effective in an earlier stage, and that the combination of chemotherapy and immunotherapy is much more effective. Considering that a durable response is achieved in most patients with complete or partial remission among stage IV patients, a durable response may be achieved at a high probability in stage III patients with an MPR after chemotherapy + immunotherapy. Furthermore, a study indicated that, among stage IV patients, PD-1 antibody therapy was more effective in those with a smaller tumor volume. In stage III patients, there is no remote metastasis, and the tumor volume may be smaller than in stage IV patients. Therefore, considering a high MPR rate after stage II/III preoperative therapy and a more favorable patient status with a small tumor volume and a small number of metastatic organs in stage III patients, chemotherapy + immunotherapy may be more effective than chemotherapy + Pembrolizumab in stage IV patients.

Based on the above background, we hypothesized that Pembrolizumab + chemotherapy might exhibit sufficient therapeutic effects similar to those of CRT in the absence of radiotherapy if PD-L1 is ≥50% in patients with non-resectable stage III non-small cell lung cancer. Furthermore, the toxicity of CRT can be avoided, and there may be a marked improvement in tolerability. Therefore, we designed a phase II, multicenter, cooperative, single-group, physician-guided trial of combination chemotherapy with Pembrolizumab and a platinum preparation in the absence of radiotherapy involving PD-L1 ≥50% stage III locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC
2. PD-L1 Total Proportion Score (TPS) ≥50%
3. Locally advanced NSCLC (unresectable stage III with indication of curative CRT based on Tumour, Node and Metastasis (TNM) classification of Union for International Cancer Control (UICC) version 8)
4. Treatment naïve for primary disease
5. Have at least measurable disease based on RECIST 1.1.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Have adequate organ function as defined in the following:

   Adequate Organ Function and Laboratory Values

   Hematological:

   Absolute neutrophil count (ANC) ≥1500/μL Platelets ≥100 000/μL Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (a)

   Renal:

   Creatinine OR Measured or calculated (b) creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × Upper Limit of Normal (ULN) OR ≥45 mL/min for participant with creatinine levels >1.5 × institutional ULN

   Hepatic:

   Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN Aspartate aminotransferase (AST) (SGOT) and Alanine transaminase (ALT) (SGPT) ≤2.5 × ULN

   Coagulation:

   International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

   Thyroid functions:

   Thyroid-Stimulating Hormone (TSH) Within institutional ULN (If TSH is not within ULN at baseline, the participant may still be eligible if T3 and free T4 are within ULN.)
   1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
   2. Creatinine clearance (CrCl) should be calculated per institutional standard.
8. Male/female participants who are at least 20 years of age on the day of signing informed consent
9. Male participants:

   A male participant must agree to use a contraception as detailed in of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

   Female participants:

   A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) as defined in OR b.) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
10. The participant is discussed in a conference including radiation oncologists.
11. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., Cytotoxic T Lymphocyte-associated Antigen 4 (CTLA-4), OX-40, CD137).
3. Has received any prior systemic anti-cancer therapy. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history of tissue/organ transplantation.
13. Has a known history of Human Immunodeficiency Virus (HIV).
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV) (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
15. Has a known history of active Tuberculosis (TB).
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | 2 years after enrollment of final patient
  Number of non-progression cases/all enrolled cases at 2 years

SECONDARY OUTCOMES:
Response rate | 6 months after enrollment of final patient
  According to RECIST
PFS | 2 years after enrollment of final patient
  According to Kaplan meier curve
OS | 2 years after enrollment of final patient
  According to Kaplan meier curve
Adverse events | 6 months and 2 years after enrollment of final patient
  Analysis of grade and incidence of adverse events

OTHER OUTCOMES:
EFFICACY assessed by Response rate in percent according to PD-L1 Total Proportion Score in percent | 6 months after enrollment of final patient
  Differences of Response rate in percent according to PD-L1 Total Proportion Score in percent
EFFICACY assessed Progression-free survival in months according to PD-L1 Total Proportion Score in percent | 2 years after enrollment of final patient
  Differences of Progression-free survival in months according to PD-L1 Total Proportion Score in percent
EFFICACY assessed by Overall survival in months according to PD-L1 Total Proportion Score in percent | 2 years after enrollment of final patient
  Differences of Overall survival in months according to PD-L1 Total Proportion Score in percent

CONTACTS AND LOCATIONS:
Overall Officials: Akito Hata, Principal Investigator — Kobe Minimally Invasive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Result] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Result] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Result] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Result] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Result] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Result] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Result] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Result] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Result] Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, Linsley PS, Thompson CB, Riley JL. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol. 2005 Nov;25(21):9543-53. doi: 10.1128/MCB.25.21.9543-9553.2005. PMID 16227604
- [Result] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Result] Yamamoto N, Nakagawa K, Nishimura Y, Tsujino K, Satouchi M, Kudo S, Hida T, Kawahara M, Takeda K, Katakami N, Sawa T, Yokota S, Seto T, Imamura F, Saka H, Iwamoto Y, Semba H, Chiba Y, Uejima H, Fukuoka M. Phase III study comparing second- and third-generation regimens with concurrent thoracic radiotherapy in patients with unresectable stage III non-small-cell lung cancer: West Japan Thoracic Oncology Group WJTOG0105. J Clin Oncol. 2010 Aug 10;28(23):3739-45. doi: 10.1200/JCO.2009.24.5050. Epub 2010 Jul 12. PMID 20625120
- [Result] Segawa Y, Kiura K, Takigawa N, Kamei H, Harita S, Hiraki S, Watanabe Y, Sugimoto K, Shibayama T, Yonei T, Ueoka H, Takemoto M, Kanazawa S, Takata I, Nogami N, Hotta K, Hiraki A, Tabata M, Matsuo K, Tanimoto M. Phase III trial comparing docetaxel and cisplatin combination chemotherapy with mitomycin, vindesine, and cisplatin combination chemotherapy with concurrent thoracic radiotherapy in locally advanced non-small-cell lung cancer: OLCSG 0007. J Clin Oncol. 2010 Jul 10;28(20):3299-306. doi: 10.1200/JCO.2009.24.7577. Epub 2010 Jun 7. PMID 20530281
- [Result] Sasaki T, Seto T, Yamanaka T, Kunitake N, Shimizu J, Kodaira T, Nishio M, Kozuka T, Takahashi T, Harada H, Yoshimura N, Tsutsumi S, Kitajima H, Kataoka M, Ichinose Y, Nakagawa K, Nishimura Y, Yamamoto N, Nakanishi Y. A randomised phase II trial of S-1 plus cisplatin versus vinorelbine plus cisplatin with concurrent thoracic radiotherapy for unresectable, locally advanced non-small cell lung cancer: WJOG5008L. Br J Cancer. 2018 Sep;119(6):675-682. doi: 10.1038/s41416-018-0243-2. Epub 2018 Sep 12. PMID 30206369
- [Result] Akamatsu H, Mori K, Naito T, Imai H, Ono A, Shukuya T, Taira T, Kenmotsu H, Murakami H, Endo M, Harada H, Takahashi T, Yamamoto N. Progression-free survival at 2 years is a reliable surrogate marker for the 5-year survival rate in patients with locally advanced non-small cell lung cancer treated with chemoradiotherapy. BMC Cancer. 2014 Jan 14;14:18. doi: 10.1186/1471-2407-14-18. PMID 24422706
- [Result] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Result] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Result] Langer CJ, Gadgeel SM, Borghaei H, Papadimitrakopoulou VA, Patnaik A, Powell SF, Gentzler RD, Martins RG, Stevenson JP, Jalal SI, Panwalkar A, Yang JC, Gubens M, Sequist LV, Awad MM, Fiore J, Ge Y, Raftopoulos H, Gandhi L; KEYNOTE-021 investigators. Carboplatin and pemetrexed with or without pembrolizumab for advanced, non-squamous non-small-cell lung cancer: a randomised, phase 2 cohort of the open-label KEYNOTE-021 study. Lancet Oncol. 2016 Nov;17(11):1497-1508. doi: 10.1016/S1470-2045(16)30498-3. Epub 2016 Oct 10. PMID 27745820
- [Result] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Result] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Result] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Result] Shu CA, Grigg C, Chiuzan C, et al. Neoadjuvant atezolizumab + chemotherapy in resectable non-small cell lung cancer (NSCLC). J Clin Oncol. 2018; 36: 15_suppl.8532
- [Result] Provencio M, Nadal E, Insa A, et al. Phase II study of neo-adjuvant chemo/immunotherapy for resectable stages IIIa non-small cell lung cancer-NADIM study-SLCG. J Thorac Oncol 2018; 13: S320.
- [Result] Tachihara M, Negoro S, Inoue T, Tamiya M, Akazawa Y, Uenami T, Urata Y, Hattori Y, Hata A, Katakami N, Yokota S. Efficacy of anti-PD-1/PD-L1 antibodies after discontinuation due to adverse events in non-small cell lung cancer patients (HANSHIN 0316). BMC Cancer. 2018 Oct 3;18(1):946. doi: 10.1186/s12885-018-4819-2. PMID 30285770
- [Result] Gettinger S, Horn L, Jackman D, Spigel D, Antonia S, Hellmann M, Powderly J, Heist R, Sequist LV, Smith DC, Leming P, Geese WJ, Yoon D, Li A, Brahmer J. Five-Year Follow-Up of Nivolumab in Previously Treated Advanced Non-Small-Cell Lung Cancer: Results From the CA209-003 Study. J Clin Oncol. 2018 Jun 10;36(17):1675-1684. doi: 10.1200/JCO.2017.77.0412. Epub 2018 Mar 23. PMID 29570421
- [Result] Huang AC, Postow MA, Orlowski RJ, Mick R, Bengsch B, Manne S, Xu W, Harmon S, Giles JR, Wenz B, Adamow M, Kuk D, Panageas KS, Carrera C, Wong P, Quagliarello F, Wubbenhorst B, D'Andrea K, Pauken KE, Herati RS, Staupe RP, Schenkel JM, McGettigan S, Kothari S, George SM, Vonderheide RH, Amaravadi RK, Karakousis GC, Schuchter LM, Xu X, Nathanson KL, Wolchok JD, Gangadhar TC, Wherry EJ. T-cell invigoration to tumour burden ratio associated with anti-PD-1 response. Nature. 2017 May 4;545(7652):60-65. doi: 10.1038/nature22079. Epub 2017 Apr 10. PMID 28397821
- [Result] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Derived] Hata A, Ninomaru T, Okada H, Kogure Y, Oki M, Katakami N, Kijima T, Yokoyama T, Matsumoto H, Sato Y, Kato T, Sugawara S, Sawada T, Yoshimura K, Seto T, Nakagawa K, Okamoto I, Yamamoto N; West Japan Oncology Group. Radiotherapy-free pembrolizumab combined with chemotherapy for locally advanced non-small-cell lung cancer with PD-L1 tumour proportion score of 50% or higher (Evolution trial): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2025 Nov;26(11):1432-1442. doi: 10.1016/S1470-2045(25)00462-0. Epub 2025 Oct 11. PMID 41082893